CLINICAL TRIAL: NCT00328445
Title: The Positive Action Program: Outcomes and Mediators
Brief Title: Randomized Trial of the Positive Action Program in Hawaii Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Principal Investigator, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA013474 (NIH)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2014-09

CONDITIONS: Character; Violence; Substance Use; Pro-social Behavior; Academic Achievement
Keywords: Curriculum; Classroom management; School-wide climate; Parent involvement
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Business as usual
- Treatment (Experimental): Positive Action
  Interventions: Behavioral: Positive Action

INTERVENTIONS:
Behavioral: Positive Action — See publications
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine the effectiveness of the Positive Action program on reducing negative behaviors, increasing positive behaviors and improving academic achievement of elementary school students.

DETAILED DESCRIPTION:
This project will: 1) evaluate the efficacy of a comprehensive, multi-grade, multi-year program, the Positive Action program (PA) designed to reduce student problem behaviors (including drug use and violence), disciplinary referrals and suspensions, and academic underachievement; 2) evaluate the effects of the program on the presumed/theoretical mediator variables; and 3) assess which of these changes in mediator variables actually mediate the effects of the program on behavior and school performance. The Hawaiian school district has agreed to implement a randomized trial of the PA program. We randomly assigned schools to PA or control conditions from strata matched on multiple indicators of risk. PA schools will receive the full PA program for four years (the 2002-03 through 2005-06 school years). This includes all materials for all students (at all grades), families, teachers, and principal, plus community kits; training for teachers and other interested staff; and continuous technical support and monitoring by a PA staff person. Data on behavior and academic achievement will be obtained from school archival records for all students for all years and, where appropriate for several years prior to the study. Students in grades 1 and 3 in the 2001-02 school year and their parents and teachers will also be followed through the project with surveys every year. The subject population will contain equal portions of males and females, and proportionate numbers of the major ethnic groups on Oahu (Hawaiian or part-Hawaiian, white, Asian, Other). Analyses will test for program effects on all hypothesized mediating variables and outcomes, and the hypothesized mediational pathways.

ELIGIBILITY:
Inclusion Criteria:

* Public elementary schools K-5 or K-6
* All students in the study cohorts

Exclusion Criteria:

* Schools performing in top 50%

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2001-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Self-reported attitudes and behaviors | 2001-2006
Teacher reports of behaviors | 2001-2006
Parent reports of student behaviors | 2001-2006

SECONDARY OUTCOMES:
School-level academic achievement test scores | 2000-2007
School-level reports of disciplinary referrals | 2000-2007
School-level reports of school quality | 2000-2007

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Flay, D.Phil., Principal Investigator — Oregon State University
Locations (3):
- United States (3):
  - Positive Action, Inc., Twin Falls, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - Oregon State University, Corvallis, Oregon

REFERENCES:
- [Background] Beets MW, Flay BR, Vuchinich S, Acock AC, Li KK, Allred C. School climate and teachers' beliefs and attitudes associated with implementation of the positive action program: a diffusion of innovations model. Prev Sci. 2008 Dec;9(4):264-75. doi: 10.1007/s11121-008-0100-2. Epub 2008 Sep 9. PMID 18780182
- [Result] Beets MW, Flay BR, Vuchinich S, Snyder FJ, Acock A, Li KK, Burns K, Washburn IJ, Durlak J. Use of a social and character development program to prevent substance use, violent behaviors, and sexual activity among elementary-school students in Hawaii. Am J Public Health. 2009 Aug;99(8):1438-45. doi: 10.2105/AJPH.2008.142919. Epub 2009 Jun 18. PMID 19542037
- [Result] Snyder F, Flay B, Vuchinich S, Acock A, Washburn I, Beets M, Li KK. Impact of a social-emotional and character development program on school-level indicators of academic achievement, absenteeism, and disciplinary outcomes: A matched-pair, cluster randomized, controlled trial. J Res Educ Eff. 2010 Jan;3(1):26-55. doi: 10.1080/19345740903353436. PMID 20414477
- [Result] Snyder FJ, Vuchinich S, Acock A, Washburn IJ, Flay BR. Improving elementary school quality through the use of a social-emotional and character development program: a matched-pair, cluster-randomized, controlled trial in Hawai'i. J Sch Health. 2012 Jan;82(1):11-20. doi: 10.1111/j.1746-1561.2011.00662.x. PMID 22142170
- See also: Link to information about the Positive Action program — http://www.positiveaction.net